CLINICAL TRIAL: NCT01113918
Title: A Study of Clinical Presentation and Cardiovascular Disease of Hyperandrogenism and Polycystic Ovary Syndrome in Obese and Non-obese Taiwanese Women
Brief Title: Expression of CVD and HA Between Obesity and Non-obesity Polycystic Ovary Syndrome (PCOS) Women in Taiwan
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Attending Doctor, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-PCOS-97070
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Obesity,; PCOS,; HA,; CVD
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obsity PCOS Women: Polycystic ovary syndrome (PCOS) was diagnosed according to the European Society for Human Reproduction (ESHRE)/American Society of Reproductive Medicine (ASRM) case definition which requires presentation of signs and/or symptoms of a minimum of 2 of the following 3 criteria: polycystic ovary morphology (PCOM), oligomenorrhea or amenorrhea (Oligo-An), androgen excess (HA).
  Body mass index (BMI) was defined as body weight in kilograms divided by body height in meters squared (kg/m2). Obesity was defined as BMI≥25 kg/m2, according to the Asia-Pacific definition.
- Non-obesity PCOS Women: The subjects BMI were less than ≥25 kg/m2 and out of criteria of PCOS by European Society for Human Reproduction (ESHRE)/American Society of Reproductive Medicine (ASRM).

SUMMARY:
Polycystic Ovarian Syndrome (PCOS) is the most common endocrine disorder in reproductive women. It is estimated that 5 to 10% of women of reproductive age have PCOS. One of the major diagnostic criteria of PCOS was chronic anovulation which lead to irregular menstruation, amenorrhea, and infertility; the other diagnostic criteria was hyperandrogenism which lead to hirsutism, acne and alopecia. Furthermore, PCOS is thought as a metabolic disorder, the long-term consequence of PCOS were diabetes mellitus and cardiovascular disease, which are potentially dangerous in women health. Early diagnosis and prevention is very important to the PCOS patients.

Obesity is the most potential risk of threat to health of populations. There is a major impact of obesity on the PCOS related disorders. Insulin resistance and distribution of adipose tissue were thought to be the important risk factors of cardiovascular and metabolic syndrome. To treat PCOS patients properly,Wan-Fang hospital had established a specific medical team. We recently published in "Fertility and Sterility" about the clinical presentation of androgen excess in Taiwanese women. Hirsutism is much less prevalence (30%) in Taiwanese PCOS women than that previous reported (65-80%) in theWestern women. It is important to know that some clinical presentation of PCOS might have ethic variance. Insulin resistance was reported as another candidate that might have ethic variance.We had reported about 40% women in PCOS women were obese, it is similar with previous literature reported. Obesity is a major factor that could be controlled during the treatment of PCOS.Weight reduction is one of our methods in PCOS treatment. The progressive results for obese PCOS women would be facing the risks of diabetes and metabolic syndrome.We thought like to evaluate the benefit of weight reduction program to the prognosis of obese women with PCOS.

Furthermore, it is known that Endothelial progenitor cells (EPC) be an early marker of cardiovascular disease, we would like to know the role of EPC to predict metabolic syndrome in women with PCOS. Wan-Fang hospital has a professional team in PCOS treatment and research which including gynecological endocrinologist, cardiologist, medical endocrinologist, specialist in weight reduction. This team had been working well for more that 4 years.

We hope we can make a contribution to the study and treatment of PCOS in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* women who had visited the Reproductive Endocrinology Clinic at Taipei Medical University - Wan Fang Medical Center during April 2004 - March 2007 with the chief complaints of menstrual irregularities, infertility, acne/or hirsutism.

Exclusion Criteria:

* women who had been diagnosed with androgen-secreting tumors.
* girls who had their menarche less than 3 years prior to the study, or who older than 40.
* women with inadequate clinical/biochemical records.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Polycystic Ovarian Syndrome(PCOS) women in wanfang hospital.
Sampling Method: Probability Sample
Enrollment: 627 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Obese | Who had visited the Reproductive Endocrinology Clinic at Taipei Medical University-Wan Fang Medical Center during April 2004 - March 2007.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taipei, Taiwan